CLINICAL TRIAL: NCT03073343
Title: A Prospective, Randomized, Open Label Trial of Two Doses of Oral Betaine in Patients With Non-alcoholic Fatty Liver Disease (NAFLD) and Elevated Alanine Aminotransferase (ALT)
Brief Title: A Prospective, Randomized, Open Label Trial of Two Doses of Oral Betaine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Timothy Morgan, MD, Chief, Hepatology, Southern California Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Betaine 2
Record Dates: First submitted 2017-02-20; First posted 2017-03-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Insulin Dependent Diabetes; ALT
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Betaine

STUDY DESIGN:
Intervention Model Description: Two cohorts of patients will be studied: Cohort 1 (diabetic) will consist of patients with a clinical diagnosis of non-insulin dependent type II diabetes mellitus; Cohort 2 (non-diabetics) will consist of patients without a clinical diagnosis of type 2 diabetes mellitus. 24 patients will be enrolled in each cohort (total of 48 patients enrolled in the study) with an anticipated drop out of 4 subjects per cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diabetic patients with NAFLD (Active Comparator): Patients will be prescribed 4 grams of betaine/day (2 grams PO BID) for the first 4 weeks of the study. After 4 weeks, patients in each cohort will be randomized (1:1) to continue receiving betaine 4 grams per day or increase to 8 grams per day for an additional 8 weeks.
  Interventions: Dietary Supplement: Betaine (trimethyglycine)
- non-diabetics with NAFLD (Active Comparator): Patients will be prescribed 4 grams of betaine/day (2 grams PO BID) for the first 4 weeks of the study. After 4 weeks, patients in each cohort will be randomized (1:1) to continue receiving betaine 4 grams per day or increase to 8 grams per day for an additional 8 weeks.
  Interventions: Dietary Supplement: Betaine (trimethyglycine)

INTERVENTIONS:
Dietary Supplement: Betaine (trimethyglycine) — Betaine (trimethyglycine) is a food supplement that is approved for sale in the United States without a prescription. In this study, betaine will be provided to patients as a powder that can be mixed with aqueous solutions and consumed orally.

SUMMARY:
Betaine (trimethyglycine) is a food supplement that is approved for sale in the United States without a prescription. In this study, betaine will be provided to patients as a powder that can be mixed with aqueous solutions and consumed orally.

DETAILED DESCRIPTION:
This is a prospective, unblinded, randomized study of oral betaine in diabetic and non-diabetic patients who have a clinical diagnosis of NAFLD and an ALT≥ 50 IU/mL. A clinical diagnosis of NAFLD is based on the presence of risk factors for NAFLD (such as overweight and insulin resistance) and the exclusion of other causes of liver disease, such as alcohol or viral hepatitis.

Two cohorts of patients will be studied: Cohort 1 (diabetic) will consist of patients with a clinical diagnosis of non-insulin dependent type II diabetes mellitus; Cohort 2 (non-diabetics) will consist of patients without a clinical diagnosis of type 2 diabetes mellitus. 24 patients will be enrolled in each cohort (total of 48 patients enrolled in the study) with an anticipated drop out of 4 subjects per cohort.

Patients will be given dietary instructions and advice on exercise appropriate for the management of NAFLD (NIDDK and liverfoundation.org handouts). Patients will be prescribed 4 grams of betaine/day (2 grams PO BID) for the first 4 weeks of the study. After 4 weeks, patients in each cohort (NIDDM and non-diabetic) will be randomized (1:1) to continue receiving betaine 4 grams per day or increase to 8 grams per day for an additional 8 weeks. All patients will be seen in clinic on a monthly basis during treatment, and again 4 and 12 weeks after completion of betaine treatment. The total duration of the study is 24 weeks (12 weeks of betaine treatment and 12 weeks of follow-up).

The primary outcome is change in ALT during 12 weeks of betaine treatment (i.e., ALT at week 12 compared with ALT at baseline (entry). Secondary outcomes include safety, efficacy of betaine in each cohort, and are changes in laboratory tests related to NAFLD.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for all patients:

1. Age 18-75 years
2. A clinical diagnosis of non-alcoholic fatty liver disease.
3. Alanine aminotransferase (ALT) levels ≥60 IU/mL
4. Laboratory tests as defined below:

   * Platelets > 100,000/dL
   * Total bilirubin < 2 mg/dL
   * Creatinine < 1.6 mg/dL

     * Inclusion Criteria for Group 1: diabetic patients

1. At least one of the following:

* Fasting blood sugar ≥ 126mg/dL
* Hemoglobin A1c (HgA1c) of > 6.5%
* 2-hour plasma glucose level of > 200mg/dL during a glucose tolerance test
* Receiving treatment with insulin sensitizing drugs (metformin) or sulfonylureas (glipizide, etc.) 3. Inclusion Criteria for Group 2: Non-diabetic patients with insulin resistance (must have both)
* Fasting blood glucose of 100-125 mg/dL and
* Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) score >3.0

Exclusion Criteria:

1. Evidence of liver disease other than non-alcoholic fatty liver disease or non-alcoholic steatohepatitis
2. Alcohol consumption of more than 12g/d (1 drink) for females or more than 24g/day (2 drinks) for males, for 3 months during the past year
3. Active substance abuse within the past year
4. Prior or ongoing use of injectable insulin
5. Use of oral corticosteroids within the prior 30 days
6. Hospitalization within the past 14 days
7. Known HIV infection
8. HgA1c >10%
9. Known heart failure of New York Heart Association class 2, 3, or 4
10. Any condition, which in the opinion of the investigator, would impede compliance or hinder the completion of the study
11. History of allergic reactions attributed to compounds of similar chemical or biologic composition to betaine
12. Current use of betaine or S-adenosylmethionine supplements, or refusal to abstain from their use during the study
13. Known cystathionine beta-synthase (CBS) deficiency.
14. Pregnancy or refusal to use birth control measures or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-11-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in alanine aminotransferase (ALT) level in all study participants | after 12 weeks of Betaine
  Compare the week 12 ALT levels with the baseline ALT in study patients. Comparison will be performed using a paired t-test.

SECONDARY OUTCOMES:
Compare changes in alanine aminotransferase (ALT) level in both cohorts | after 12 weeks of Betaine
  A Paired T test analysis will compare changes in ALT levels between Patients with NIDDM (cohort 1) and Patients without NIDDM (cohort 2)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Morgan, MD, Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with anyone outside authorized research personnel.

REFERENCES:
- [Background] Matteoni CA, Younossi ZM, Gramlich T, Boparai N, Liu YC, McCullough AJ. Nonalcoholic fatty liver disease: a spectrum of clinical and pathological severity. Gastroenterology. 1999 Jun;116(6):1413-9. doi: 10.1016/s0016-5085(99)70506-8. PMID 10348825
- [Background] Caldwell SH, Oelsner DH, Iezzoni JC, Hespenheide EE, Battle EH, Driscoll CJ. Cryptogenic cirrhosis: clinical characterization and risk factors for underlying disease. Hepatology. 1999 Mar;29(3):664-9. doi: 10.1002/hep.510290347. PMID 10051466